CLINICAL TRIAL: NCT03516786
Title: Quality of Recovery After Quadratus Lumborum Block for Cesarean Section: A Prospective Pilot Study
Brief Title: Quality of Recovery After Quadratus Lumborum Block for Cesarean Section.
Status: Completed | Type: Observational
Sponsor: Corniche Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ch1712171
Record Dates: First submitted 2018-03-19; First posted 2018-05-04 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective study is to evaluate the recovery after cesarean section in patients who will receive Quadratus Lumborum Block (QLB) as a part of multimodal analgesia using Postoperative quality of recovery scale.

DETAILED DESCRIPTION:
Several researchers had evaluated the effectiveness of QLB in controlling postoperative pain in different patient populations. In these studies, the effectiveness of the QLB was mainly assessed by postoperative pain scores and analgesia consumption, rather than adapting any of the more comprehensive recovery scales .

Postoperative quality of recovery scale (PostopQRS) is a relatively new recovery score, which was first published on 2010, and was designed to be a tool for assessment of multiple domains in recovery. In this assessment tool, recovery was defined as return to the pre-surgery base line scores or better.

The aim of this prospective study is to evaluate the recovery after cesarean section in patients who will receive Quadratus Lumborum Block QLB as a part of multimodal analgesia using Postoperative quality of recovery scale.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) physical status II, normal singleton pregnancy, 37 weeks gestation or more Scheduled for elective cesarean section

Exclusion Criteria:

* Patients refusing spinal
* Patients with BMI >35 kg/m2).
* Expected difficult surgery (> 3 previous sections, abnormal placentation, prolonged surgery more than 2 hours from skin to end) and Estimated Blood Loss more than 1500).
* Expected difficult spinal anesthesia.
* Abnormal coagulation and other contraindications for spinal anesthesia and/or QLB
* Patient with chronic pain.
* Patient treated from psychosis.
* Patients with communication, language barriers .

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women at term
Study Population: Twenty five parturients, with American Society of Anesthesiologists (ASA) physical status II, with normal singleton pregnancy, at 37 weeks gestation or more, admitted to Corniche Hospital for elective caesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
change from baseline postoperative quality of recovery score | 72 hours
  Domains of postoperative recovery score are :
  1. The physiologic domain .
  2. The nociceptive domain
  3. The emotive domain .
  4. Activities of daily living
  5. Cognitive domain
  6. Over all patients perspective domain

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, Principal Investigator — Corniche Hospital; Amr Maher, MD, Principal Investigator — Corncihe hospital
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates